CLINICAL TRIAL: NCT03672396
Title: Feasibility Study of a Home-Based Exercise Intervention Program for Patients With Metastatic Castration-Resistant Prostate Cancer Receiving Androgen Deprivation Therapy (ADT)
Brief Title: Home-based Exercise Intervention for Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC1613
Record Dates: First submitted 2018-08-31; First posted 2018-09-14 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2020-12

CONDITIONS: Castration-resistant Prostate Cancer; Androgen Deprivation Therapy
Keywords: exercise; hormone therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Single-arm study with ~30 men being recruited and 20-25 who complete all aspects of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based Exercise (Experimental): The sole intervention group will complete a combination of aerobic and strength training ~3 times per week for 12 weeks with each session lasting 1 hour.
  Interventions: Behavioral: Home-based exercise

INTERVENTIONS:
Behavioral: Home-based exercise — The intervention consists of aerobic and strength training ~3 times per week for 12 weeks with each session lasting 1 hour. The progressive aerobic exercise will involve walking that varies from from 15 to 30 minutes done 2-4 times per week at an intensity from 40% to 65% of heart rate reserve. Therabands elastic bands will be used to perform 12 to 15 repetitions per exercise. Once a participant can comfortably complete 15 repetitions for all prescribed sets, they will increase resistance by moving up to the next band. The training volume increased from 1 set per exercise on week 1 to 3 sets by week 12.

SUMMARY:
This single arm, multi-site pilot study aims to evaluate the feasibility of recruiting and adherence to a 12 week home-based exercise intervention to be conducted in men with metastatic castration resistant prostate cancer (mCRPC) receiving androgen deprivation therapy (ADT). Thirty patients will be enrolled, with the expectation that 20-25 will complete all follow-up measures.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the feasibility and adherence to a home-based 12 week exercise intervention in mCRPC patients receiving ADT. It will also examine if a home-based exercise intervention can improve muscle strength, body composition, physical function, cardiopulmonary function fatigue, and patient reported outcomes (fatigue, depression, quality of life (QoL)).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease that has progressed despite castrate levels of testosterone (surgically or medically castrated, with testosterone levels of < 50 ng/dL) receiving ADT. This will be verified by assessing total testosterone levels within 4 weeks prior to enrollment.
* No current chemotherapy.
* Patients may be receiving additional hormonal therapy agents including but not limited to antiandrogens (e.g. bicalutamide, enzalutamide) and CYP17 inhibitors (e.g. abiraterone).
* Ability to engage safely in moderate exercise as determined by their treating physician.
* Not previously engaged in regular exercise training (<3 or more d/wk for > 30 min/d or <90 mins per week total including strength training, aerobic training, or walking) in the past 6 months.
* Access to a computer or a smart phone for syncing and uploading wearable activity data.
* Be able to speak and read English.

Exclusion Criteria:

* Any condition that causes severe pain with exertion.
* History of bone fractures.
* Active cardiovascular disease including any of the following:

  * New York Heart Association (NYHA) Grade II or greater congestive heart failure .
  * History of myocardial infarction or unstable angina within 6 months prior to Day 1.
  * History of stroke or transient ischemic attack within 6 months prior to Day 1.
* Acute or chronic respiratory disease that is severe enough to compromise the ability of the participant to safely engage in exercise training protocol.
* Acute or chronic bone/joint/muscular abnormalities compromising their ability to exercise.
* Neurological conditions that affect balance and, or muscle strength.
* Dementia, altered mental status or any psychiatric condition prohibiting the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik D Hanson, PhD, Principal Investigator — UNC-Chapel Hill
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Comprehensive Cancer Center, Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
Both sites (UNC and WF) are adding and storing data on a secure, centralized server. No individual data will be made available to protect the identity of the patients in the trial.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4/16/2017 through 12/5/2019 from referrals from medical oncologists from three institutions.
Pre-assignment Details: 62 subjects were referred to the study. Of this, 40 did not participate or qualify for the study. 22 subjects were consented and 16 completed all aspects of the trial.
Period: Overall Study
Arm/Group | Home-based Exercise
Started | 22
Completed | 16
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Data were reported only on those subjects who completed the intervention and performed testing at baseline and post intervention.
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Height [Mean (Standard Deviation); unit: cm] | 172.4 (4.6)
Mass [Mean (Standard Deviation); unit: kg] | 86.2 (19.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.90 (6.00)
Duration of Androgen Deprivation Therapy (ADT) [Mean (Standard Deviation); unit: days] | 1132 (1369)
Previous Prostatectomy [Count of Participants; unit: Participants] | 7
Previous Radiotherapy [Count of Participants; unit: Participants] | 11
Previous Chemotherapy [Count of Participants; unit: Participants] | 5
Time since Chemotherapy [Mean (Standard Deviation); unit: months] | 13 (5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Complete the Pre/Post Exercise Intervention Testing.
Description: To estimate the feasibility of a 12 week, home-based exercise intervention in metastatic castrate resistant prostate cancer (mCPRC) patients undergoing androgen deprivation therapy by reporting the percentage of patients who complete the pre/post testing following the intervention.
  This was calculated as the number of subjects who completed the trial compared to the total number who completed baseline testing.
Time Frame: 12 weeks after baseline testing
Population: All participants in the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 22
Participants | 16

2. Secondary Outcome: Adherence to the Intervention
Description: To report the level of adherence to the exercise intervention in patients completing pre/post testing. Successful adherence to the program is completion of 75% of all prescribed exercise and will be assessed using wearable technology to track walking and exercise logs to track resistance training adherence.
  Adherence was determined as the number of exercise sessions attempted/completed over the total number of session prescribed.
Time Frame: 12 weeks after baseline testing
Population: This analysis was restricted to subjects who completed the intervention and returned their training logs.
Measure: Number; unit: percentage of total sessions prescribed
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 14
percentage of total sessions prescribed
  Overall | 80.1
  Walking | 65.5
  Resistance Training | 72.8

3. Secondary Outcome: Physical Function: 6m Walk
Description: The time to complete (in sec) the 6m rapid walk test will be performed.
Time Frame: 12 weeks after baseline testing
Population: Data from pre vs. post intervention were analyzed using a paired t-test only in subjects who completed all aspects of the trial.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 16
seconds
  Baseline | 4.4 (1.5)
  Post Intervention | 4.5 (1.5)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — Paired t-test analysis between baseline and post-testing values from a single group of individuals who completed both testing sessions; p = 0.378, t-test, 2 sided; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.2 to 0.4]

4. Secondary Outcome: Physical Function: Timed Up and Go
Description: The time to complete (in sec) the 2.44m (8 ft) timed up and go test will be performed as an indicator of agility, balance, and physical function. A lower total time is indicative of greater performance.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 16
seconds
  Baseline | 10.4 (9.1)
  Post Intervention | 10.8 (11.0)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.586, t-test, 2 sided; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-1.0 to 1.7]

5. Secondary Outcome: Physical Function: Stair Climb
Description: The time to climb a flight of stairs (in sec) will be performed as an indicator of functional strength, muscle power, and balance. A lower total time (and higher calculated power output) is indicative of greater performance.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 16
seconds
  Baseline | 6.4 (2.8)
  Post Intervention | 6.2 (3.2)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.252, t-test, 2 sided; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.7 to 0.2]

6. Secondary Outcome: Physical Function: 400m Walk
Description: The time to walk 400m (in sec) will be performed as an indicator of walking endurance and gait speed will be determined. A lower total time and higher gait speed indicates greater cardiorespiratory capacity and will be correlated with cardiopulmonary function scores (outcome 14).
Time Frame: 12 weeks after baseline testing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 15
seconds
  Baseline | 329.8 (97.8)
  Post Intervention | 313.5 (87.3)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.111, t-test, 2 sided; Mean difference calculated as Post - Pre; Mean Difference (Final Values) = -16.3, 95% CI 2-sided [-36.9 to 4.3]

7. Secondary Outcome: Patient Reported Outcomes: Fatigue
Description: Fatigue will be measure using the Functional Assessment of Chronic Illness Therapy Fatigue, a 1 page form that uses a rating scale that goes from 0 to 52. It assesses the patient's fatigue levels in the last 7 days. It also measures how usual activities, performing work, walking, relationship, and enjoyment of life are affected by fatigue. A higher score indicates higher quality of life (and lower fatigue).
Time Frame: 12 weeks after baseline testing
Population: Data from pre vs. post intervention were analyzed using a paired t-test only in subjects who completed all aspects of the trial and returned the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 9
score on a scale
  Baseline | 39 (10)
  Post Intervention | 40 (11)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.579, t-test, 2 sided; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-4.3 to 7.2]

8. Secondary Outcome: Patient Reported Outcomes: Quality of Life
Description: Quality of life will be measured using the Functional Assessment of Cancer Therapy-Prostate (FACT-P). The FACT-P is composed of both multi-item scales and single-item measures. These include physical, social, emotional, and functional well-being, along with an assessment of prostate-specific health status. five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the individual questions are scored from 0-4 with total scores ranging between 0 and 156 where a higher number represents higher QoL.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 9
score on a scale
  Baseline | 119 (20)
  Post Intervention | 119 (16)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.948, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-3.9 to 3.7]

9. Secondary Outcome: Patient Reported Outcomes: Depression
Description: Depression will be measured using the Hospital Anxiety and Depression Scale, a concise, self-administered 1 page form that categorizes anxiety and depression. The total score goes from 0-21, and scores are categorized from minimal to severe depression/anxiety. Higher total scores indicate greater levels of depression.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 9
score on a scale
  Baseline | 3 (2)
  Post Intervention | 3 (3)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.594, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.1 to 0.7]

10. Secondary Outcome: Patient Reported Outcomes: Anxiety
Description: as for outcome 9
Time Frame: 12 weeks after baseline testing
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 9
score on a scale
  Baseline | 4 (3)
  Post Intervention | 3 (2)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.274, t-test, 2 sided; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.3 to 0.7]

11. Secondary Outcome: Muscle Size (Cross-sectional Area)
Description: Muscle size will be analyzed using ultrasound of the vastus lateralis of the dominant leg. All assessments will be completed before and after the intervention to determine the muscle size. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality.
Time Frame: 12 weeks after baseline testing
Population: Data from pre vs. post intervention were analyzed using a paired t-test only in subjects who completed all aspects of the trial and were tested at the University of North Carolina (UNC) site only. Equipment to perform this analysis at the Wake Forest site was not available.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 13
cm^2
  Baseline | 8.3 (2.9)
  Post Intervention | 10.2 (4.0)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.013, t-test, 2 sided; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [0.48 to 3.29]

12. Secondary Outcome: Muscle Quality
Description: Muscle architecture will be analyzed using ultrasound of the vastus lateralis of the dominant leg. All assessments will be completed before and after the intervention to determine the muscle quality. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality. Muscle quality is reported in arbitrary units, where a lower value indicates a higher/better muscle quality.
Time Frame: 12 weeks after baseline testing
Population: Data from pre vs. post intervention were analyzed using a paired t-test only in subjects who completed all aspects of the trial and were tested at the UNC site.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 13
unitless
  Baseline | 110.2 (22)
  Post Intervention | 114.3 (16.6)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.369, t-test, 2 sided; Mean Difference (Final Values) = 4.16, 95% CI 2-sided [-5.54 to 13.85]

13. Secondary Outcome: Chest Press Maximal Strength
Description: Upper and lower body muscle strength will be assessed using the chest and leg presses. Maximal strength is defined as the highest load (kilograms) that the participant can successfully lift one time. Greater maximal strength is associated with greater physical function and QoL.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 14
kg
  Baseline | 62.4 (21.4)
  Post Intervention | 62.0 (13.3)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.945, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-13.5 to 12.7]

14. Secondary Outcome: Chest Press Muscle Endurance
Description: Upper and lower body muscle endurance will be assessed using the chest and leg presses. Muscle endurance is the total number of repetitions completed using 70% of maximal load determined during muscle strength testing (outcome 12). Greater muscle endurance are associated with greater physical function and QoL.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: number of repetitions completed
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 14
number of repetitions completed
  Baseline | 14.1 (5)
  Post Intervention | 15.4 (6.8)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.420, t-test, 2 sided; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.0 to 4.6]

15. Secondary Outcome: Leg Press Maximal Strength
Description: as for outcome 13
Time Frame: 12 weeks after baseline testing
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 14
kg
  Baseline | 142.1 (49.1)
  Post Intervention | 141.5 (52.0)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.941, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-16.9 to 15.8]

16. Secondary Outcome: Leg Press Muscle Endurance
Description: as for outcome 14
Time Frame: 12 weeks after baseline testing
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: number of repetitions completed
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 12
number of repetitions completed
  Baseline | 11.8 (6.7)
  Post Intervention | 14.1 (6.4)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.203, t-test, 2 sided; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-1.4 to 5.9]

17. Secondary Outcome: Cardiopulmonary Function
Description: To report changes in cardiopulmonary function following the intervention. Cardiopulmonary function (VO2 peak) will be assessed using a graded exercise test on a treadmill. Patients will begin the test walking slowly on the treadmill and every two minutes, the grade and speed of the treadmill will be increased in a progressive manner until fatigue occurs. Respiratory gases will be collected throughout the test and analyzed using a metabolic cart to determine oxygen utilization and carbon dioxide production. The maximal oxygen uptake that is recorded will be used as a marker of aerobic fitness.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 15
mL/kg/min
  Baseline | 19.3 (4.0)
  Post Intervention | 20.1 (5.6)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.057, t-test, 2 sided; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.04 to 2.6]

18. Secondary Outcome: Lean Mass
Description: To report changes in total lean mass following the intervention. Total body lean mass will be measured using dual-energy x-ray absorptiometry (DXA) before and after the intervention.
Time Frame: 12 weeks after baseline testing
Population: Data from pre vs. post intervention were analyzed using a paired t-test only in subjects who completed all aspects of the trial and the body composition scans.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 15
kg
  Baseline | 54.5 (8.6)
  Post Intervention | 51.4 (16)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.809, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.0 to 1.3]

19. Secondary Outcome: Fat Mass
Description: To report changes in total fat mass following the intervention. Total fat mass will be measured using dual-energy x-ray absorptiometry (DXA) before and after the intervention.
Time Frame: 12 weeks after baseline testing
Population: Data from pre vs. post intervention were analyzed using a paired t-test only in subjects who completed all aspects of the trial and completed the body composition scans.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 15
kg
  Baseline | 30 (12.9)
  Post Intervention | 28.4 (15.2)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.191, t-test, 2 sided; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.3 to 1.1]

20. Secondary Outcome: Percent Body Fat
Description: To report changes in relative fat mass following the intervention. Total body percent fat (percentage of fat mass relative to total mass) will be measured using dual-energy x-ray absorptiometry (DXA) before and after the intervention.
Time Frame: 12 weeks after baseline testing
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percentage of total body mass
Arm/Group | Home-based Exercise
Number analyzed (Participants) | 15
percentage of total body mass
  Baseline | 34.0 (6.1)
  Post Intervention | 34.3 (6.6)
Statistical Analysis 1: Comparison: Home-based Exercise; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.237, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.3 to 1.3]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Home-based Exercise
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-based Exercise (N=22)
calcium pyrophosphate deposition disease (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03672396/Prot_SAP_000.pdf